CLINICAL TRIAL: NCT04281173
Title: Evaluation of Multifocal ERG and Visual Field Changes After Vitrectomy and ILM Peeling
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Almoatz bellah zohier Mohammed, director, Assiut University
Other Study IDs: ERG in ILM peeling
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evulate changes in MfERG, VF and OCT after viterctomy associated with ILM peeling.

DETAILED DESCRIPTION:
Macular epiretinal membrane (ERM) is a disorder of the vitreomacular interface characterized by ﬁbrocellular proliferation on the anterior surface of the internal limiting membrane (ILM) of the macula. Pars plana vitrectomy with ERM removal and inner limiting membrane peeling is the standard surgical treatment for an ERM. ILM peeling is performed to eliminate the scaffold for myoﬁbroblast proliferation and any microscopic ERM in order to prevent ERM recurrence. ILM peeling is indicated for other pathologies other than ERM such as, diabetic macular edema, and macular hole. ILM peeling is a traumatic procedure that may have many effects on the underlying inner retinal layers that may lead to changes in retinal function.

Retinal edema, eccentric scotoma, dissociation of the nerve fiber layer, iatrogenic punctuate chorioretinopathy, and subretinal, retinal, and vitreous hemorrhage are well described secondary to the surgical trauma of peeling in addition to stain toxicity. Investigation of these changes may assist in aiding the development of minimally traumatic techniques for ILM removal .

Evaluation of functional changes may include visual field and Multifocal electroretinography assessment. Visual field defect after vitrectomy a well known post operative complication usually in eyes that underwent fluid air exchange, the cause of visual field defect remain unclear.

Optical Coherence Tomography (OCT), imaging is done to evaluate inner retinal layers after ILM peeling,High myopic eyes might develop more severe, "scattered" inner retinal defects after ILM peeling.

Multifocal electroretinography (mfERG), has been used to assess visual function and the electrophysiologic responses of multiple retinal locations of the macular area

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic ERM,
2. Primary full thickness macular hole,
3. Lamellar macular hole, and
4. Vitromacular traction

Exclusion Criteria:

* 1-Patients with a secondary ERM,

  1. diabetic retinopathy,
  2. venous occlusion,
  3. retinal detachment,
  4. uveitis, and
  5. trauma. 2-Other ocular pathologies that could interfere with the functional results

  <!-- -->

  1. dense cataract ,
  2. glaucoma, and
  3. previous retinal surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with diopathic ERM,Primary full thickness macular hole, Lamellar macular hole, and Vitromacular traction
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
BCVA | 6 months
  after ILM peeling

REFERENCES:
- [Background] Mensch G. Dental licensing. Midwest Dent. 1968 Oct;44(10):13. No abstract available. PMID 5247634